CLINICAL TRIAL: NCT00301639
Title: A PET Study Examining Pharmacokinetics and Dopamine Transporter Receptor Occupancy Of Two Long-Acting Formulations of Methylphenidate in Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: McNeil Consumer & Specialty Pharmaceuticals, a Division of McNeil-PPC, Inc. (Industry)
Responsible Party: Thomas J. Spencer, MD, Massachusetts General Hospital
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 2004-p-002189
Record Dates: First submitted 2006-03-10; First posted 2006-03-13 (Estimated); Last update posted 2011-07-12 (Estimated); Status verified 2011-07

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Methylphenidate

INTERVENTIONS:
Drug: OROS methylphenidate hydrochloride
Drug: methylphenidate hydrochloride

SUMMARY:
The specific aim of this study is to document the pharmacokinetics of dopamine transporter DAT receptor occupancy of OROS MPH and Metadate CD using PET scanning with C-11 Altropane as the ligand. We hypothesize that CNS DAT occupancy of OROS MPH will be greater than that of Metadate CD at 10 hours after administration.

DETAILED DESCRIPTION:
OROS-MPH's pharmacokinetic profile uses an increasing delivery of MPH over the day (ascending pharmacokinetic curve). It was designed to replace IR-MPH TID treatment. Another new long-acting formulation is Metadate CD. Metadate CD consists of capsules with two types of beads. It was designed to replace IR-MPH BID treatment. The main target of MPH in the brain is the dopamine transporter (DAT). We have an exquisitely sensitive methodology to measure DAT occupancy using C-11 Altropane and Positron Emission Tomography (PET). The time course of decay of the C-11 Altropane permits repeated imaging, thus allowing documentation of the pharmacokinetics of DAT receptor occupancy.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent to participate in the study.
2. Age: 18 - 55
3. If female, non-pregnant, non-nursing, using an adequate form of birth control or a negative serum pregnancy test.
4. Supine and standing blood pressure within the range 110/60 to 150/90 mmHg.
5. Heart rate, after resting for 5 minutes, within the range 46-90 beats/min.
6. Subjects who are within 20% of the ideal weight for height.
7. Right handed.

Exclusion Criteria:

1. Diagnosis of any psychotic disorder, bipolar disorder, severe depression, severe anxiety, or Autism. Subjects with mild mood, oppositional, conduct, and anxiety disorders may be permitted to participate if considered appropriate by the investigator.
2. Scores of Baseline Scales:

   Hamilton Depression Scale > 17 (out of a possible 67 on the 21-item scale) (Hamilton 1960) Beck Depression Inventory > 19 (out of a possible 63 on the 21-item scale) (Beck et al 1961) Hamilton Anxiety Scale > 21 (out of a possible 56 on the 14-item scale) (Hamilton 1959)
3. Tics or Tourette's Syndrome.
4. Diagnosis of ADHD
5. History of head trauma with loss of consciousness, organic brain disorders, seizures, or neurosurgical intervention.
6. Any clinically significant chronic medical condition, in the judgment of the investigator.
7. Mental impairment as evidenced by an I.Q. <75.
8. Exposure to dopamine receptor antagonists within the previous three (3) months.
9. Exposure to radiopharmaceuticals within four (4) weeks prior to PET scan.
10. Subjects receiving psychotropic medication.
11. Any clinically significant abnormality in the screening laboratory tests, vital signs, or 12-lead ECG, outside of normal limits.
12. Any woman of childbearing potential who is seeking to become pregnant or suspects that she may be pregnant.
13. Subjects with a known recent history (within the past six (6) months) of illicit drug or alcohol dependence.
14. Subjects diagnosed with glaucoma.
15. Subjects at risk for MPH toxicity (e.g. individuals with arrhythmias, coronary artery disease, etc.).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40
Dates: Start 2005-03; Primary Completion 2005-12 (Actual); Study Completion 2005-12

PRIMARY OUTCOMES:
The DAT receptor occupancy of OROS MPH and Metadate CD using PET scanning with C-11 Altropane. Objective measures also provided by d and l ritalinic acid and methylphenidate levels at pre-dose, hr 9, 10 and 11.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Spencer, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Cambridge, Massachusetts, United States